CLINICAL TRIAL: NCT03433313
Title: A Phase III, Randomized, Multicenter, Double-blind Study to Compare Efficacy and Safety of EG12014 With Herceptin as Neoadjuvant Treatment in Combination With Anthracycline/Paclitaxel Systemic Therapy in HER2-Positive Early Breast Cancer
Brief Title: Efficacy and Safety Study of EG12014 Compared With Herceptin in Subjects With HER2 Positive Early Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EirGenix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EGC002; 2017-003973-33 (EudraCT Number)
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EG12014 (Experimental): Epirubicin and cyclophosphamide followed by EG12014 plus paclitaxel. All patients will be scheduled for surgery (breast and axillary lymph nodes) at 3 to 6 weeks after completion of neoadjuvant chemotherapy.
  Interventions: Drug: EG12014
- Herceptin (Active Comparator): Epirubicin and cyclophosphamide followed by Herceptin plus paclitaxel. All patients will be scheduled for surgery (breast and axillary lymph nodes) at 3 to 6 weeks after completion of neoadjuvant chemotherapy.
  Interventions: Drug: Herceptin

INTERVENTIONS:
Drug: EG12014 — EG12014 6mg/kg is ongoing to be administered after 8mg/kg loading dose.
  Arms: EG12014
Drug: Herceptin — Herceptin 6mg/kg is ongoing to be administered after 8mg/kg loading dose.
  Arms: Herceptin

SUMMARY:
The purpose of this research study is to compare the efficacy and safety of EG12014 with Herceptin as neoadjuvant treatment for 12 weeks, followed by surgery and subsequent EG12014 or Herceptin adjuvant treatment for up to 12 months.

ELIGIBILITY:
1. Provide signed and dated written informed consent before entering the study. The informed consent will cover both parts of the study (neoadjuvant part and adjuvant part).
2. Female, ≥18 and ≤65 years of age.
3. Histologically-confirmed invasive carcinoma of the breast (American Joint Committee on Cancer [AJCC, vs. 8.0] Stage II, IIIa).
4. Operable breast cancer, planned surgical resection of breast tumor (mastectomy or lumpectomy) and sentinel or axillary lymph nodes.
5. Unilateral, measurable tumor of the breast >2 cm in diameter.
6. HER2 positive tumor, defined as 3+ score by IHC or fluorescence positive by FISH, as confirmed by central laboratory.
7. Known estrogen receptor (ER) and progesterone receptor (PrR) status at study entry.
8. Adequate bone marrow function, defined as granulocyte count of ≥1.500/µL, and platelet count of ≥100.000/µL.
9. Adequate hepatic and renal function, defined as:

   bilirubin within normal range

   alanine aminotransferase (ALT) ≤2 x upper limit of normal (ULN)

   aspartate aminotransferase (AST) ≤2 x ULN

   gamma glutamyl transferase (GGT) ≤3 x ULN

   serum creatinine <1.5 ULN
10. International normalized ratio ≤1.5×ULN (2 to 3×ULN if on anticoagulants) or prothrombin time ≤1.5×ULN; activated partial thromboplastin time ≤1.5×ULN.
11. Hemoglobin concentrations ≥10 g/dL.
12. Eastern Cooperative Oncology Group (ECOG) score of 0 or 1.
13. LVEF ≥55%, measured by multiple-gated acquisition (MUGA) scan or echocardiography.
14. Negative pregnancy test at entry, women of childbearing potential have to use contraceptives during the course of the study.

Females with childbearing potential must provide a negative serum pregnancy test at Screening and must be using adequate birth control. Adequate birth control is defined as agreement to consistently practice an effective and accepted method of contraception throughout the duration of the study and for 7 months after study drug treatment. These methods include hormonal contraceptives, intrauterine device, or double barrier contraception (i.e., condom + diaphragm) or a male partner with documented vasectomy.

Non-childbearing potential is defined as post-menopausal for at least 1 year or surgical sterilization or hysterectomy at least 3 months before study start.

Exclusion Criteria:

1. Bilateral breast cancer.
2. Pregnancy or lactation or considering becoming pregnant.
3. Metastases, other than sentinel/axillary lymph nodes.
4. Previous treatment (chemotherapy, biologic therapy, radiation, or surgery) for invasive malignant disease or other concomitant malignancy, other than basal cell carcinoma of the skin. Previous treatment for carcinoma in situ of the cervix is allowed.
5. Previous treatment with Herceptin.
6. Angina pectoris or arrhythmia requiring medication; poorly controlled hypertension; history of myocardial infarction or cardiac failure, New York Heart Association (NYHA) class II or higher; clinically significant cardiac valvular disease; hemodynamic effective pericardial effusion; other cardiomyopathies; LVEF of <55%.
7. Any investigational treatment less than 30 days prior to study entry, or within a time interval less than at least 5 half-lives of the investigational medicinal product, whichever is longer.
8. Positive diagnostic test for hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
9. History of hypersensitivity to drugs with similar chemical structures to trastuzumab.
10. History of, or known current problems with, drug or alcohol abuse.
11. Other serious illness, medical disorder or condition that, in the opinion of the Investigator, would make the patient unsuitable for participation in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 807 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Determination of pathologic complete response (pCR) at time of surgery | At the time of surgery (3-6 weeks after completion of neoadjuvant chemotherapy)
  pCR is defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled sentinel and/or axillary lymph nodes

SECONDARY OUTCOMES:
pCR at the time of surgery | At the time of surgery (3-6 weeks after completion of neoadjuvant chemotherapy)
  pCR is defined as the absence of residual invasive cancer and of DICS (ypT0 ypN0) from breast tissue and sentinel/axillary lymph nodes, as assessed by central laboratory
pCR at the time of surgery | At the time of surgery (3-6 weeks after completion of neoadjuvant chemotherapy)
  pCR is defined as the absence of invasive cancer in breast tissue only (ypT0/is) as assessed by central laboratory
Event-free survival (EFS) up to end of study (EOS) | Randomization to date of progression or end of study (up to approximately 24 months or death)
  EFS is defined as time from initial randomization to the date when disease recurrence or progression (local, regional, distant or contralateral) is diagnosed according to institutional standard, or date of death of any cause, whichever is earlier
Overall response (OR) prior to surgery | At screening and prior to surgery (3-6 weeks after completion of neoadjuvant chemotherapy)
  Objective response is defined as partial response (PR) or complete response (CR) according to RECIST v1.1
Overall survival (OS) up to End of Study (EOS) | Randomization to end of study (up to approximately 24 months or death)
  OS up to EOS is defined as time from the date of initial randomization to the date of death
Incidence of AEs | From time of informed consent to end of study (up to approximately 25 months or death)
  Incidence of AEs (including severity, seriousness, and relationship to study drug) and laboratory abnormalities
Evaluation of Immunogenicity of EG12014 and Herceptin | Prior to 1st infusion of study drug, during neoadjuvant treatment, after the last dose of neoadjuvant treatment, during adjuvant treatment, and End of Treatment
  Titer of anti-drug antibodies (ADA)
Measure serum trastuzumab concentration | Prior to 1st infusion of study drug, during neoadjuvant treatment after the last dose of neoadjuvant treatment, during adjuvant treatment, and End of Treatment
  Measure serum trastuzumab concentration for EG12014 and Herceptin arms

CONTACTS AND LOCATIONS:
Locations (91):
- United States (2):
  - Detroit Clinical Research Center, Farmington Hills, Michigan
  - Aultman Hospital, Cancer Center, Canton, Ohio
- Belarus (6):
  - Brest Regional Oncology Center, Brest
  - Gomel Regional Clinical Oncology Center, Homyel
  - N.N. Aleksandrov Republican Research Oncology and Medical Radiology Center, Lesnoy
  - Minsk City Clinical Oncology Center, Minsk
  - Mogilev Regional Oncology Center, Mogilev
  - Vitebsk Regional Clinical Oncology Center, Vitebsk
- Chile (2):
  - Medical Research Limited Society, Temuco
  - Oncocentro Apys, Viña del Mar
- Colombia (2):
  - Clinic Life Foundation, Medellín
  - Rodrigo Botero SAS, Medellín
- Georgia (9):
  - LTD High-Tech Hospital MedCenter, Batumi
  - JSC "Evex Hospitals, Kutaisi
  - LTD Acad. F. Todua Medical Center - LTD Research Institute of Clinical Medicine, Tbilisi
  - LTD Aversi Clinic, Tbilisi
  - LTD Cancer Research Centre, Tbilisi
  - LTD Health House, Tbilisi
  - LTD Institute of Clinical Oncology, Tbilisi
  - LTD S.Khechinashvili University Hospital, Tbilisi
  - Malkhaz Katsiashvili Multiprofile Emergency Medicine Center, Tbilisi
- India (5):
  - Cytecare Cancer Hospitals, Bengaluru
  - King George's Medical University, Department of Endocrine surgery, Shatabdi Phase II, Lucknow
  - Tata Memorial Centre, Mumbai
  - HCG NCHRI Cancer Centre, Nagpur
  - Christian Medical College, Department of Medical Oncology, Vellore
- Russia (30):
  - Arkhangelsk Clinical Oncology Center, Arkhangelsk
  - Chelyabinsk Regional Clinical Oncology and Nuclear Medicine Center, Chelyabinsk
  - Evimed, LLC, Chelyabinsk
  - Ivanovo Regional Oncology Center, Ivanovo
  - Republican Clinical Oncology Center, Kazan'
  - Krasnoyarsk A.I. Kryzhanovsky Regional Oncology Center, Krasnoyarsk
  - Kursk Regional Clinical Oncology Center, Kursk
  - N.N. Blokhin National Medical Oncology Research Center, Moscow
  - National Medical Research Center for Radiology, Moscow
  - Vitamed" LLC, Moscow
  - A.F.Tsyb Medical Radiology Research Center, Obninsk
  - Clinical Oncology Center, Omsk
  - Pyatigorsk Interdistrict Oncology Center, Pyatigorsk
  - Rostov Oncology Research Institute, Rostov-on-Don
  - Regional Clinical Oncology Center, Ryazan
  - AV Medical Group, Saint Petersburg
  - City Clinical Oncology Center, Saint Petersburg
  - Clinic "Mart", Saint Petersburg
  - I.I. Mechnikov North-Western State Medical University, Saint Petersburg
  - Leningrad Regional Oncology Center (Outpatient Department), Saint Petersburg
  - Leningrad Regional Oncology Center (Surgery Department), Saint Petersburg
  - N.N. Petrov National Medical Research Center of Oncology, Saint Petersburg
  - Oncology Center of Moskovskiy District, Saint Petersburg
  - Private Medical Institution "EVROMEDSERVIS", Department of Oncology, Saint Petersburg
  - St. Petersburg Clinical Research and Practical Center for Specialized Types of Medical Care (Oncology), Saint Petersburg
  - Republican Oncology Center, Saransk
  - Oncology Center #2, Sochi
  - Tomsk National Research Medical Center, Tomsk
  - Regional Clinical Oncology Center, Veliky Novgorod
  - Volgograd Regional Clinical Oncology Center, Volgograd
- South Africa (5):
  - GVI Oncology, Cape Gate Oncology Centre, Cape Town
  - The Oncology Centre, Durban
  - Medical Oncology Centre of Rosebank, Johannesburg
  - Little Company of Mary Medical Center, Department of Oncology, Pretoria
  - University of Pretoria, Department of Medical Oncology, Pretoria
- Keimyung University - Dongsan Medical Center, Daegu, South Korea
- Taiwan (6):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Ukraine (23):
  - Chernihiv Regional Oncology Center, Chernihiv
  - Chernivtsi Regional Clinical Oncology Center, Chernivtsi
  - Clinical Oncology Center, Dnipro
  - Dnipropetrovsk City Multispecialty Clinical Hospital #4, Department of Chemotherapy, Dnipro
  - Prikarpattia Clinical Oncology Center, Ivano-Frankivsk
  - Communal Non-profit enterprise "Regional Center of Oncology", Kharkiv
  - State Institution: S.P. Hryhoriev Institute of Medical Radiology under the Ukrainian Academy of Medical Sciences, Department of Clinical Oncology and Hematology, Kharkiv
  - Khmelnytskyi Regional Oncology Center, Khmelnytskyi
  - Kryvyi Rih Oncology Center, Department of Chemotherapy, Kryvyi Rih
  - Kyiv City clinical Hospital #2, Kyiv
  - Kyiv Regional Oncology Center, Department of Mastology, Kyiv
  - Medical Center "Verum", Kyiv
  - Medical Center of First Private Clinic, Kyiv
  - Volyn Regional Oncology Center, Department of Chemotherapy, Lutsk
  - Public Institution under Lviv Regional Council: Lviv Regional Treatment and Diagnostics Oncology Center, Department of Chemotherapy, Lviv
  - Mariupol Oncology Center, Mariupol
  - Odesa Regional Clinical Hospital, Center for Mastology, Department of Thoracic Surgery, Odesa
  - Odesa Regional Oncology Center, Odesa
  - Ternopil Regional Clinical Oncology Center, Department of Chemotherapy, Ternopil
  - Central City Clinical Hospital, Department of Oncology and Radiology, Uzhhorod
  - Zakarpattia Regional Clinical Oncology Center, Department of Chemotherapy, Uzhhorod
  - Podillia Regional Oncology Center, Vinnytsia
  - Zhytomyr Regional Oncology Center, Zhytomyr

IPD SHARING:
Plan to Share IPD: Undecided